CLINICAL TRIAL: NCT00764569
Title: a Non-invasive Device for the Detection, Diagnosis and Screening of Oral Pathology
Brief Title: The Investigation of a Fluorescence/Elastic Scattering Spectroscopy (F-ESS) Device for Oral Tissue Characterization
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Petra Wilder-Smith, DDS., PhD., Professor, Director of Dentistry, University of California, Irvine
Other Study IDs: 20086355
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Other Lesions of Oral Mucosa
Keywords: oral tissue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oral Tissue measurement: Fluorescence/Elastic Scattering Spectroscopy Oral tissue measurement
  Interventions: Device: Fluorescence/Elastic Scattering Spectroscopy

INTERVENTIONS:
Device: Fluorescence/Elastic Scattering Spectroscopy — Fluorescence/Elastic Scattering Spectroscopy Oral tissue measurement

SUMMARY:
The overall objective of this work is to identify changes in the optical properties of oral tissues to develop a non-invasive tool for the detection, diagnosis and screening of oral pathology so that treatment can be provided at the earliest possible time.

DETAILED DESCRIPTION:
Specifically, we will be obtaining optical spectroscopic data using a fiber optic contact probe that exploits elastic-scattering spectroscopy and fluorescence spectroscopy. Both of these technique have independently shown to provide signatures for the onset of cancer, with varied success. The purpose of this effort is to combine the two techniques and develop and understanding of the signatures obtained in both normal and abnormal oral tissue with simultaneous collection of these optical signatures.

ELIGIBILITY:
Inclusion Criteria:

* adult over 18 years of age

Exclusion Criteria:

* younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic Tool | 4 weeks
  Fluorescence/Elastic Scattering Spectroscopy Oral tissue measurement

CONTACTS AND LOCATIONS:
Overall Officials: Petra Wilder-Smith, DDS, PhD, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (2):
- United States (2):
  - Beckman Laser Institute Medical clinic, Irvine, California
  - UCI student health center, Irvine, California